CLINICAL TRIAL: NCT01597960
Title: Yoga And Cardiovascular Health Trial
Acronym: YACHT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 12/LO/0597
Record Dates: First submitted 2012-05-08; First posted 2012-05-15 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2012-06

CONDITIONS: Cardiovascular Disease
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Yoga 12 week programme (Active Comparator): Usual care (standard cardiac rehabilitation programme) plus yoga intervention.
  Interventions: Other: Yoga
- Usual care (No Intervention): Usual care (standard cardiac rehabilitation programme) only.

INTERVENTIONS:
Other: Yoga — Those randomised to usual care plus the yoga intervention will be required to attend yoga classes twice a week for 12 weeks alongside their cardiac rehabilitation programme. There will be 24 yoga classes in total, of which, we require the participant to attend a minimum of 18. The yoga classes will be conducted by a teacher certified in yoga and cardiac rehabilitation and will encompass physical fitness (yoga poses), stress reduction (breath control and meditation) and positive lifestyle changes (diet, smoking and alcohol).
  Arms: Yoga 12 week programme

SUMMARY:
The benefits of alternative therapeutic approaches, such as yoga, are poorly understood and this is particularly true of the beneficial effects on cardiovascular disease (CVD) risk. It is hoped that a better understanding of the value of this therapy will provide a sound scientific basis for including yoga in mainstream clinical practice. The investigators propose to study a group of 80 participants (40 Indian Asians and 40 Europeans) recruited from a cardiac rehabilitation programme in West London post-angioplasty as treatment for an acute coronary syndrome. Those who agree will undergo a series of baseline and follow-up measurements. 20 Indian Asians and 20 Europeans will be randomized to the yoga intervention plus their standard cardiac rehabilitation programme (usual care), and the remaining 20 Indian Asians and 20 Europeans will be randomized to usual care alone. Baseline and follow-up measurements will be performed on all participants. In order to determine the acute effects of yoga the group randomised to the yoga intervention will also undergo a series of acute tests before and after their first yoga session.

DETAILED DESCRIPTION:
The benefits of alternative therapeutic approaches, such as yoga, are poorly understood and this is particularly true of the beneficial effects on cardiovascular disease (CVD) risk. It is hoped that a better understanding of the value of this therapy will provide a sound scientific basis for including yoga in mainstream clinical practice. The investigators propose to study a group of 80 participants (40 Indian Asians and 40 Europeans) recruited from a cardiac rehabilitation programme in West London post-angioplasty as treatment for an acute coronary syndrome. Those who agree will undergo a series of baseline and follow-up measurements. 20 Indian Asians and 20 Europeans will be randomized to the yoga intervention plus their standard cardiac rehabilitation programme (usual care), and the remaining 20 Indian Asians and 20 Europeans will be randomized to usual care alone. Baseline and follow-up measurements will be performed on all participants; these include: Demographic & health questionnaire, Lifestyle questionnaires focusing on diet and exercise, Fasting bloods sampling (for cardiovascular risk factors and markers), Saliva sampling (x 5 samples for salivary cortisol and alpha-amylase), Anthropometrics - height, weight and waist and hip circumference, Bioimpedence - measurement of total body fat, 3D and Doppler echocardiography, Carotid IMT, Resting brachial blood pressure, Central blood pressure (tonometery at the radial artery), Pulse Wave Velocity, 12 lead ECG, Cardiopulmonary exercise testing, Combined 24hr BP & ECG monitor, Accelerometer (3 days). In order to determine the acute effects of yoga the group randomised to the yoga intervention will also undergo a series of acute tests before and after their first yoga session. These include: Exercise capacity, Saliva sampling (x 5 samples for salivary cortisol and alpha-amylase) and combined 24hr BP & ECG monitor.

ELIGIBILITY:
Inclusion Criteria:

* Aged 35-80 years.
* Male or female.
* European or Indian Asian descent.
* Able to understand English or Punjabi.
* Referred to a cardiac rehabilitation programme in West London post-angioplasty as treatment for an acute coronary syndrome.

Exclusion Criteria:

* Adults under 35 years or above 80 years.
* Adults aged 35-80 years who are not competent to give consent.
* Co-morbid disease or mobility limitations that would preclude participation in cardiac rehabilitation and our investigations.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Cardiopulmonary function | Week 0 (pre intervention) and week 12 (post intervention)
  To perform a mechanistic study that determines the acute and chronic effects of yoga on cardiopulmonary function, autonomic function, blood pressure and heart rate.

SECONDARY OUTCOMES:
Blood pressure | Week 0 (pre intervention), week 1 (pre & post 1st yoga class), and week 12 (post intervention)
  Blood pressure will be measured at baseline, at the beginning and end of the first yoga class, and immediately after the 12 week intervention.
Heart rate and heart rate variability | Week 0 (pre intervention), week 1 (pre & post 1st yoga class), and week 12 (post intervention)
  Heart rate and heart rate variability will be measured at baseline, at the beginning and end of the first yoga class, and immediately after the 12 week intervention.
Stress hormones | Week 0 (pre intervention), week 1 (pre & post 1st yoga class), and week 12 (post intervention)
  Stress hormones will be measured at baseline, at the beginning and end of the first yoga class, and immediately after the 12 week intervention.
Exercise capacity | Week 0 (pre intervention), week 1 (pre & post 1st yoga class), and week 12 (post intervention)
  Exercise capacity will be measured at baseline, at the beginning and end of the first yoga class, and immediately after the 12 week intervention.
Body fat | Week 0 (pre intervention) and week 12 (post intervention)
  Body fat will be measured at baseline and immediately after the 12 week intervention.
Glucose and lipids | Week 0 (pre intervention) and week 12 (post intervention)
  Glucose and lipids will be measured at baseline and immediately after the 12 week intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Nishi Chaturvedi, Principal Investigator — Imperial College London
Locations (1):
- International Centre for Circulatory Health, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Tillin T, Tuson C, Sowa B, Chattopadhyay K, Sattar N, Welsh P, Roberts I, Ebrahim S, Kinra S, Hughes A, Chaturvedi N. Yoga and Cardiovascular Health Trial (YACHT): a UK-based randomised mechanistic study of a yoga intervention plus usual care versus usual care alone following an acute coronary event. BMJ Open. 2019 Nov 3;9(11):e030119. doi: 10.1136/bmjopen-2019-030119. PMID 31685500